CLINICAL TRIAL: NCT03094234
Title: 8mm-TIPS Versus Endoscopic Variceal Ligation (EVL) Plus Propranolol for Prevention of Variceal Rebleeding in Patients With Child A Cirrhosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, Principal Investigator, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8mm-TIPS-ChildA
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Propranolol

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8mm-TIPS (Active Comparator): Patients in this group would underwent TIPS placement with 8mm-diameter ePTFE-covered stents.
  Interventions: Device: 8mm-TIPS
- EVL plus propranolol (Active Comparator): Patients in this group would underwent sequential endoscopic variceal ligation and propranolol treatment.
  Interventions: Procedure: endoscopic variceal ligation (EVL); Drug: Propranolol

INTERVENTIONS:
Device: 8mm-TIPS — Patients in this group would underwent TIPS placement with 8mm-diameter ePTFE-covered stents.
  Arms: 8mm-TIPS
Procedure: endoscopic variceal ligation (EVL) — Patients in this group would underwent sequential endoscopic variceal ligation and propranolol treatment.
  Arms: EVL plus propranolol
Drug: Propranolol — Appropriate dose of propranolol was administered to the patients.
  Arms: EVL plus propranolol

SUMMARY:
The aim of this study was to conduct a prospective randomized trial to compare TIPS with 8mm expanded polytetrafluoroethylene(ePTFE)-covered stents and endoscopic variceal ligation plus propranolol for the prevention of recurrent esophageal variceal bleeding in patients with Child A cirrhosis

DETAILED DESCRIPTION:
For the prevention of recurrent esophageal variceal bleeding, previous clinical studies and meta-analysis show that patients treated with transjugular intrahepatic portosystemic shunt (TIPS) have lower rebleeding rates compared with endoscopic therapy. However, TIPS is associated with higher rates of portosystemic encephalopathy and does not show survival benefit. TIPS with a small-diameter may achieve sufficient portal decompression and reduce the incidence of hepatic encephalopathy. The aim of this study was to conduct a prospective randomized trial to compare TIPS with 8mm ePTFE-covered stents and endoscopic variceal ligation plus propranolol for the prevention of recurrent esophageal variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

Cirrhosis Patients who had bled from esophageal varices (≥5days and ≤28days) Child-Pugh A -

Exclusion Criteria:

The presence of gastric varices Non-cirrhotic portal hypertension Portal vein thrombosis The history of hepatic encephalopathy Total bilirubin ≥51.3 umol/L Previous treatment of TIPS or surgery Proven malignancy including hepatocellular carcinoma Contraindications to TIPS、EVL or propranolol End-stage renal disease under renal replacement therapy; Cardiorespiratory failure Pregnancy or patients not giving informed consent for endoscopic procedure

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2022-03-28 (Estimated); Study Completion 2022-03-28 (Estimated)

PRIMARY OUTCOMES:
Variceal rebleeding rate | 3 years
  Analysis

SECONDARY OUTCOMES:
Hepatic encephalopathy rate | 3 years
  Analysis
TIPS dysfunction rate | 3 years
  Analysis
The incidence of complications | 3 years
  Analysis
Mortality rate | 3 years
  Analysis

CONTACTS AND LOCATIONS:
Locations (1):
- West china hospital, Chengdu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Simonetti RG, Perricone G, Robbins HL, Battula NR, Weickert MO, Sutton R, Khan S. Portosystemic shunts versus endoscopic intervention with or without medical treatment for prevention of rebleeding in people with cirrhosis. Cochrane Database Syst Rev. 2020 Oct 22;10(10):CD000553. doi: 10.1002/14651858.CD000553.pub3. PMID 33089892